CLINICAL TRIAL: NCT01308918
Title: The New GlideRite DLT Stylet®: An Observational Study
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean Bussières, Professeur de clinique, Laval University
Other Study IDs: IUCPQ-20420
Record Dates: First submitted 2011-03-01; First posted 2011-03-04 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-02

CONDITIONS: Double Lumen Tube Intubation
Keywords: Thoracic surgery; Double lumen tube intubation; GlideScope; Stylet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GlideScope DLT intubation: Patients having a thoracic surgery (non cardiac) via either thoracoscopy or thoracostomy. Patients were all 18 years old or over, and have read, understood and signed an informed consent at the preoperative evaluation or on surgery morning.

SUMMARY:
Thoracic surgeries usually require lung isolation techniques. Double-lumen tube (DLT), either right or left sided, is the most frequent tool used to realize this technique. In front of difficult airways, the use of videolaryngoscopy (GllideScope®) (GS) may advantageous. Hypothesis: We will test the hypothesis that under GS, the use of a specific semi-rigid stylet is efficacious to insert a DLT, and also safe. The increased rigidity of the GlideRite DLT Stylet for double-lumen tubes will enable the DLT to keep its form while it is railroaded into superior airways. This new stylet combined to Glidescope® utilization will increase the rate of successful intubation, especially in patients with difficult airways. This technique will allow us to directly intubate with a DLT using the GlideScope®, avoiding a beforehand SLT intubation and airway exchange catheter use. Consequently, its use could reduce risks associated to blind insertion of DLT with airway exchange catheter (airway traumatism and pulmonary aspiration). Primary objective: To determine the GlideRite DLT Stylet efficiency for double-lumen tubes orotracheal intubation under videolaryngoscopy (GllideScope®). Secondary objectives: to time successful intubation, to count the number of intubation attempt, to verify the influence of difficult intubation score (DIS) on successful intubation, and to log complications associated to its use. Exclusion criterion are: previous history of difficult intubation, anticipated difficult mask ventilation, and anticipated difficult intubation. Conclusion: The aim of using the GlideRite DLT Stylet for an orotracheal intubation under videolaryngoscopy is to allow the primary intubation with a DLT in patients with abnormal superior airways. These anomalies are more and more frequent. Alternative airway management implies more manipulations, leading to an increased risk of oxygen desaturation, lung aspiration, and airway lesions. Moreover, these alternatives take more time than using a Glidescope, which can be compare to direct laryngoscopy. The development of a semi-rigid stylet, such as the GlideRite DLT Stylet, is a great advancement in the management of primary intubation with DLT, mainly in face of difficult airways.

DETAILED DESCRIPTION:
INTRODUCTION Anesthesia in thoracic surgery (non cardiac) often requires pulmonary isolation techniques in order to facilitate the surgery, to protect a healthy lung, and to control the ventilation. The double lumen tube (DLT), in right and left version, is the technique of choice to obtain lung isolation, whereas the bronchial blocker can also be used.

Double-lumen tube One-lung ventilation is required in most of thoracic surgeries. Many strategies can be used to achieve lung isolation: 1) use of endobronchial tube, 2) use of a single-lumen tube (SLT) and a bronchial blocker (BB),or 3) use of a double-lumen tube (DLT). There is many advantages of using a DLT: easier to position, shorter time of lung collapsing and re-expansion than BB, each lung can be suctioned/ventilated separately, and less subject to displacement than BB. Since no medical instrument is perfect, DLT has also some inconvenient: DLT are larger, and less compliant than a SLT. They also have two cuffs, one bronchial and another one tracheal. The latter is causing problem when intubating patients with teeth at the superior jaw. Precautions have to be taken to avoid rupturing the tracheal cuff. These characteristics are exaggerated when anesthesiologist faces a patient with a difficult airway. These cases are usually managed by first proceeding to a standard intubation with a SLT, second, use an airway exchange catheter (AEC) to withdraw the SLT, and then, advance the DLT into the proper position. Thereafter, the gold standard is to confirm the DLT position with a fiberoptic bronchoscope (FOB). If direct laryngoscopy provides poor glottis visualization, another option is to proceed to a FOB-assisted DLT intubation.

Video laryngoscopes Over the last decade, video laryngoscopes have been developed to handle difficult airway management. They have the advantage of improving Cormack-Lehane (CL) grade over direct laryncoscopy. Many manufacturers distribute video laryngoscopes: the Storz® C-MAC™, the McGrath® Series-5™, and the GlideScope® Video Laryngoscope™ (GVL) are few examples. This latter is frequently used in our centre to allow tracheal intubation with a SLT in numerous situations where conventional laryngoscopy is not possible. The GVL requires the same technique than a direct laryngoscopy without a line of sight, turning CL Grade III or IV into CL Grade I or II.

Stylet To facilitate the endotracheal tube (ETT) insertion using the GVL, either a semi-rigid or a malleable stylet must be used. There is also a lot of discussion about the best stylet configuration allowing the tip of the ETT to be positioned at the glottis opening and advancing the tube into the trachea, but no consensus has been obtained yet. Difficult airway management may be optimized by shaping the SLT using a malleable stylet, directing the ETT through vocal cords. The main problem of malleable stylet is that it loses its initial shape when the ETT goes through narrow airways. It is why many clinicians prefer the semi-rigid stylet when using the GlideScope®. Double-lumen tubes are already supplied with a malleable aluminum stylet in order for them to maintain their initial shape, and some authors found that accuracy of placement have improved when it is retained into a left-DLT for the entire intubation procedure.

New semi-rigid stylet Video laryngoscopes have been designed to be mostly used with SLT, but recent publications have suggested using a GlideScope® for primary DLT placement in difficult airways, as described by Hernandez, A et al. in 2005 and Chen, A et al. in 2008. Even if DLT are provided with a stylet, the technique of intubation with the GVL remains difficult, mainly because the aluminum stylet is too malleable. Verathon Inc. has marketed the GlideRite® rigid stylet, especially design to use with the GlideScope®. Its length fits most of SLT, its shape is adapted to the GVL's curvature, and the curvature can be modified to accommodate a difficult airway only with intentional movement. In collaboration with Verathon Inc., we have designed a new semi-rigid intubating stylet that can be use for primary DLT intubation with the Glidescope® Videolaryngoscope, the GlideRite DLT Stylet®. This improved intubating tool is sharing the same curve but is longer than the GlideRite® rigid stylet. It present a specific handle to fit with the DLT and to orient the distal extremity into the right or left bronchus. The new stylet fits 35 to 41 French, left of right-sided DLTs. Anticipated benefits of this new design are a shorter time required to position the DLT, less intubating attempt, lower risk of trauma to the airway, lower risk of desaturation and, lower risk of tracheal cuff' rupture, resulting in a one-step lung isolation.

HYPOTHESIS We believe that, under video laryngoscopy, the use of the semi-rigid GlideRite DLT Stylet® for primary insertion of DLT is possible.

The gain of rigidity that we have developed for the GlideRite DLT Stylet® imposes its shape to the DLT, and conserves it while the tube is guided through the superior airway. We hope that the combination of both the GlideScope® and the new semi-rigid stylet will increase the number of successful primary intubation with a double lumen tube. Furthermore, its utilization could drastically decrease associated risks of blind DLT intubation with an AEC. These risks are oxygen desaturation, pulmonary aspiration, and superior airway trauma.

OBJECTIVES The primary objective of this observational study is to determine the GlideRite DLT Stylet® efficiency during endotracheal intubation with a double lumen tube under video laryngoscopy (GlideScope®).

The secondary objectives are:

1. To time the intubating process.
2. To count the number of attempt to obtain a successful intubation.
3. To verify the correlation between the difficult intubation score and a successful intubation.
4. To note all complications associated to the GlideRite DLT Stylet® utilization.

METHODS After obtaining local REB approval, 50 patients having a thoracic surgery (non cardiac) via either thoracoscopy or thoracostomy, were enrolled to this observational study between May 14th 2010 and January 17th 2011.

Intraoperative proceeding Before anesthesia was induced, patients were pre-oxygenated in order to obtain an inspired-expired O2 gradient ≤10%. Anesthesia was performed in conformity with local practice standards. Curarization was achieved by injecting a dose of ≥1.0 mg/kg (ideal body weight) of rocuronium (Zémuron®, Merck & Co., Whitehouse Station, NJ, USA). If mask ventilation was proven to be difficult, the patient was excluded from the study. The malleable stylet was removed from the DLT (Broncho-Cath R- or L-DLT, 35 to 41Fr, Mallinckrodt Inc, St-Louis, MO, USA) and replaced with a GlideRite DLT Stylet® (Verathon Medical ULC, Burnaby, BC, Canada). Before proceeding to the intubation, curarization level was verified with a neuromuscular stimulator, absence of thumb movement when a train-of-four was applied allowed us to begin the protocol.

The timer was started when either the GlideScope® blade (Verathon Medical ULC, Burnaby, BC, Canada) was inserted between the lips and stopped when the tracheal cuff was passed through the vocal cords. In case of patients presenting with upper teeth, the timer was started when the DLT was inserted between the lips. Immediately after intubation, intratracheal position was confirmed with FOB. When a patient had teeth at the superior jaw, the DLT was inserted first into the mouth in order to avoid rupturing the tracheal cuff. External larynx manipulations were allowed at all time. If after one (1) minute, the intubation was not successful, the anesthesiologist could then modify the stylet shape. If after two (2) minutes, the intubation was still not achieved, the DLT and GVL blade were withdrawn, and mask ventilation was started again. At that time, the anesthesiologist could use the intubation technique of his choice. The position of the DLT was confirmed by the visualization of the trachea through the FOB. Throughout this process, if oxygen saturation dropped below 94%, mask ventilation was started to increase saturation up to 98% or more before another intubation could be attempted. If oxygen saturation dropped below 90%, mask ventilation was started to increase saturation up to 98% or more, the patient was then excluded from the study, and the anesthesiologist could use the intubation technique of his choice.

Statistical analysis Data obtained during the preoperative period will be correlated with the success rate, the time to achieve a successful intubation and, the number of attempt.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Elective thoracic surgery (non cardiac)

Exclusion Criteria:

* history of a difficult intubation in the past
* anticipated difficult mask ventilation
* anticipated difficult intubation according to the anesthesiologist's evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients having an elective thoracic surgery (non cardiac) via either thoracopscopy or thoracostomy. Patients were all 18 years old or over, and have read, understood and signed an informed consent at the preoperative evaluation or on surgery morning.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean S Bussières, MD, Principal Investigator — Laval University
Locations (1):
- Institut de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Background] Aps C, Towey RM. Experiences with fibre-optic bronchoscopic positioning of single-lumen endobronchial tubes. Anaesthesia. 1981 Apr;36(4):415-8. doi: 10.1111/j.1365-2044.1981.tb10250.x. No abstract available. PMID 7246992
- [Background] Campos JH. An update on bronchial blockers during lung separation techniques in adults. Anesth Analg. 2003 Nov;97(5):1266-1274. doi: 10.1213/01.ANE.0000085301.87286.59. PMID 14570636
- [Background] Cohen E. Recommendations for airway control and difficult airway management in thoracic anesthesia and lung separation procedures. Are we ready for the challenge? Minerva Anestesiol. 2009 Jan-Feb;75(1-2):3-5. Epub 2008 Nov 28. No abstract available. PMID 19039300
- [Background] Brodsky JB. Lung separation and the difficult airway. Br J Anaesth. 2009 Dec;103 Suppl 1:i66-75. doi: 10.1093/bja/aep262. PMID 20007992
- [Background] Fortier G, St-Onge S, Bussieres J. Two other simple methods to protect the tracheal cuff of a double-lumen tube. Anesth Analg. 1999 Oct;89(4):1064. doi: 10.1097/00000539-199910000-00047. No abstract available. PMID 10512293
- [Background] Perlin DI, Hannallah MS. Double-lumen tube placement in a patient with a difficult airway. J Cardiothorac Vasc Anesth. 1996 Oct;10(6):787-8. doi: 10.1016/S1053-0770(96)80208-4. No abstract available. PMID 8910162
- [Background] Cooper RM. Use of a new videolaryngoscope (GlideScope) in the management of a difficult airway. Can J Anaesth. 2003 Jun-Jul;50(6):611-3. doi: 10.1007/BF03018651. PMID 12826557
- [Background] Rope TC, Loughnan BA, Vaughan DJ. Videolaryngoscopy--an answer to difficult laryngoscopy? Eur J Anaesthesiol. 2008 May;25(5):434-5. doi: 10.1017/S0265021507002931. No abstract available. PMID 18377671
- [Background] Turkstra TP, Harle CC, Armstrong KP, Armstrong PM, Cherry RA, Hoogstra J, Jones PM. The GlideScope-specific rigid stylet and standard malleable stylet are equally effective for GlideScope use. Can J Anaesth. 2007 Nov;54(11):891-6. doi: 10.1007/BF03026792. PMID 17975233
- [Background] Neustein SM. The GlideScope-specific rigid stylet to facilitate tracheal intubation with the Glidescope. Can J Anaesth. 2008 Mar;55(3):196-7; author reply 197. doi: 10.1007/BF03016103. No abstract available. PMID 18310639
- [Background] van Zundert A, Maassen R, Lee R, Willems R, Timmerman M, Siemonsma M, Buise M, Wiepking M. A Macintosh laryngoscope blade for videolaryngoscopy reduces stylet use in patients with normal airways. Anesth Analg. 2009 Sep;109(3):825-31. doi: 10.1213/ane.0b013e3181ae39db. PMID 19690253
- [Background] Maassen R, Lee R, Hermans B, Marcus M, van Zundert A. A comparison of three videolaryngoscopes: the Macintosh laryngoscope blade reduces, but does not replace, routine stylet use for intubation in morbidly obese patients. Anesth Analg. 2009 Nov;109(5):1560-5. doi: 10.1213/ANE.0b013e3181b7303a. Epub 2009 Aug 27. PMID 19713258
- [Background] Dupanovic M, Diachun CA, Isaacson SA, Layer D. Intubation with the GlideScope videolaryngoscope using the "gear stick technique". Can J Anaesth. 2006 Feb;53(2):213-4. doi: 10.1007/BF03021834. No abstract available. PMID 16434769
- [Background] Muallem M, Baraka A. Tracheal intubation using the GlideScope with a combined curved pipe stylet, and endotracheal tube introducer. Can J Anaesth. 2007 Jan;54(1):77-8. doi: 10.1007/BF03021905. No abstract available. PMID 17197473
- [Background] Jones PM, Turkstra TP, Armstrong KP, Armstrong PM, Cherry RA, Hoogstra J, Harle CC. Effect of stylet angulation and endotracheal tube camber on time to intubation with the GlideScope. Can J Anaesth. 2007 Jan;54(1):21-7. doi: 10.1007/BF03021895. PMID 17197464
- [Background] Dow WA, Parsons DG. 'Reverse loading' to facilitate Glidescope intubation. Can J Anaesth. 2007 Feb;54(2):161-2. doi: 10.1007/BF03022022. No abstract available. PMID 17272262
- [Background] Cuchillo JV, Rodriguez MA. Considerations aimed at facilitating the use of the new GlideScope videolaryngoscope. Can J Anaesth. 2005 Jun-Jul;52(6):661; author reply 661-2. doi: 10.1007/BF03015790. No abstract available. PMID 15983166
- [Background] Lieberman D, Littleford J, Horan T, Unruh H. Placement of left double-lumen endobronchial tubes with or without a stylet. Can J Anaesth. 1996 Mar;43(3):238-42. doi: 10.1007/BF03011741. PMID 8829862
- [Background] Hernandez AA, Wong DH. Using a Glidescope for intubation with a double lumen endotracheal tube. Can J Anaesth. 2005 Jun-Jul;52(6):658-9. doi: 10.1007/BF03015787. No abstract available. PMID 15983163
- [Background] Chen A, Lai HY, Lin PC, Chen TY, Shyr MH. GlideScope-assisted double-lumen endobronchial tube placement in a patient with an unanticipated difficult airway. J Cardiothorac Vasc Anesth. 2008 Feb;22(1):170-2. doi: 10.1053/j.jvca.2007.04.006. Epub 2007 Jun 27. No abstract available. PMID 18249357
- [Background] Weller RM. Gum elastic bougie for difficult double-lumen intubation. Anaesthesia. 1998 Mar;53(3):311. No abstract available. PMID 9613285
- [Background] Hagihira S, Takashina M, Taenaka N, Yoshiya I. Placement of double-lumen tubes with a stylet. Can J Anaesth. 1997 Jan;44(1):101. doi: 10.1007/BF03014336. No abstract available. PMID 8988836
- [Background] Thomas V, Neustein SM. Tracheal laceration after the use of an airway exchange catheter for double-lumen tube placement. J Cardiothorac Vasc Anesth. 2007 Oct;21(5):718-9. doi: 10.1053/j.jvca.2006.08.002. Epub 2006 Nov 30. No abstract available. PMID 17905282

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 14th 2010 and January 17th 2011, 50 patients were enrolled in the study at the end of their pre-operative visit to the thoracic surgery department.
Pre-assignment Details: No enrolled participant were excluded from the study. All participants were included into the same group.
Groups:
- GlideScope DLT Intubation With GlideRite DLT Stylet: The double lumen tube (DLT) is the technique of choice to obtain lung isolation. The GlideScope® (GLS, video laryngoscope allowing vizualisation of the airway and tube placement, has been used with a high level of success to assist positioning a single lumen tube (SLT) in normal situations and mainly in situations where the airway is considered or proven to be difficult.We have designed a new semi-rigid intubating stylet, the GlideRite DLT Stylet® (GR-DLT-S), which can be used for primary DLT intubation with the GLS. This pilot study was planned to observe the efficiency and the safety of the GR-DLT-S for primary insertion of DLT with the GLS in patients presenting a normal superior airway. After obtaining local IRB approval, 50 patients scheduled for thoracic surgery (non cardiac) via either thoracoscopy or thoracostomy at l'Institut de cardiologie et de pneumologie de Québec, were enrolled in this observational study.
Period: Overall Study
Arm/Group | GlideScope DLT Intubation With GlideRite DLT Stylet
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GlideScope DLT Intubation
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 58.7 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Region of Enrollment [Number; unit: participants]
  Canada | 50
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 26.8 (4.8)
Weight [Mean (Standard Deviation); unit: kg] | 74.3 (14.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Successfull Primary Placement of the Double Lumen Tube.
Description: To evaluate the number of participants where GlideRite DLT Stylet® associated to the video laryngoscopy (GlideScope®)allowed the primary placement of the double lumen tube into their trachea.
Time Frame: 1 hour (Post intubation)
Measure: Number; unit: Participants
Arm/Group | GlideScope DLT Intubation
Number analyzed (Participants) | 50
Participants | 49

2. Secondary Outcome: Duration of the Intubating Process
Description: The timer was started when the GLS blade was inserted between the lips and stopped when the proximal part of the tracheal cuff was passed through the vocal cords. When a patient had teeth at the superior jaw, the DLT was first inserted into the mouth prior to the insertion of the GLS blade in order to avoid rupturing the tracheal cuff. For these cases, the timer was started when the DLT was inserted between the lips.
Time Frame: 1 hour (Post intubation)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GlideScope DLT Intubation
Number analyzed (Participants) | 50
Seconds | 46.3 (32.3)

3. Secondary Outcome: Number of Attempt to Obtain a Successful Intubation
Time Frame: 1 hour (Post intubation)
Measure: Number; unit: Attempts
Arm/Group | GlideScope DLT Intubation
Number analyzed (Participants) | 50
Attempts
  One (1) attempt | 37
  Two (2) attempts | 11
  Three (3) attempts | 1
  Failure | 1

4. Secondary Outcome: Correlation Between the Difficult Intubation Score and a Successful Intubation
Time Frame: 1 hour (Post intubation)
Reporting Status: Not Posted
Measure: Least Squares Mean; unit: participants

5. Secondary Outcome: Number of Complications Associated to the GlideRite DLT Stylet® Utilization
Description: Complications defined either as oxygen desaturation below 95%, oxygen desaturation below 90%, minor bleeding, anatomic lesion.
Time Frame: 1 hour (Post intubation)
Measure: Number; unit: Participants
Arm/Group | GlideScope DLT Intubation
Number analyzed (Participants) | 50
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the moment the intubation process began until the double lumen tube was secured in place. (about 15 minutes).
Description: "0" means that no serious adverse event was noted throughout the entire study.
Arm/Group | GlideScope DLT Intubation
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No